CLINICAL TRIAL: NCT00803296
Title: The Impact of Obesity and Insulin Resistance on the Incretin Effect in Patients With Type 2 Diabetes and Healthy Subjects
Brief Title: Incretin Effect in Lean and Obese Subjects
Acronym: BMI-INK
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Dr. Filip K. Knop, MD PhD, University Hospital, Gentofte, Copenhagen
Other Study IDs: BMI-INK
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2008-12

CONDITIONS: Incretin Effect; Insulin Resistance; Type 2 Diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Obese patients with type 2 diabetes: Patients with type 2 diabetes and BMI>33
  Interventions: Other: Oral glucose tolerance test (OGTT); Other: Isoglycemic intravenous glucose infusion
- Obese subjects with normal glucose tolerance: Subjects with normal glucose tolerance and BMI>33
  Interventions: Other: Oral glucose tolerance test (OGTT); Other: Isoglycemic intravenous glucose infusion
- Lean subjects with type 2 diabetes: Patients with type 2 diabetes and BM<25
  Interventions: Other: Oral glucose tolerance test (OGTT); Other: Isoglycemic intravenous glucose infusion
- Lean subjects with normal glucose tolerance: Subjects with normal glucose tolerance and BM<25
  Interventions: Other: Oral glucose tolerance test (OGTT); Other: Isoglycemic intravenous glucose infusion

INTERVENTIONS:
Other: Oral glucose tolerance test (OGTT)
Other: Isoglycemic intravenous glucose infusion

SUMMARY:
The incretin effect is markedly reduced in patients with type 2 diabetes. Data support the notion that this deficiency is a consequence of the diabetic state. However, the impact of insulin resistance on the incretin effect in obese individuals who uphold a normal glucose tolerance (NGT) despite their insulin resistant state remains to be elucidated. The primary aim of the present study is to evaluate the separate impact of one of the cornerstones of type 2 diabetic pathophysiology, namely insulin resistance, on the incretin effect in lean and obese patients with type 2 diabetes and in two matched normal-glucose tolerant groups of healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 3 months
* Normal blood hemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease
* Diabetic nephropathy
* Treatment with medication that can not be stopped for 12 hours

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lean and obese patients with type 2 diabetes; and matched healthy control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Incretin effect | 2 days

SECONDARY OUTCOMES:
Insulin resistance | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Tina Vilsbøll, MD DMSc, Study Chair — Department of Internal Medicine F, Gentofte Hospital, University of Copenhagen
Locations (1):
- Gentofte Hospital, University of Copenhagen, Hellerup, Copenhagen, Denmark